CLINICAL TRIAL: NCT04814069
Title: A Multicenter Phase II Trial of Post-operative Concurrent Chemoradiotherapy Using Weekly Cisplatin With Tislelizumab for Patients With High-risk Head and Neck Squamous Cell Carcinoma：The POTENTIAL Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Guopei Zhu, Dr., Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021HNRT01
Record Dates: First submitted 2021-03-23; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Head and Neck Cancer; Radiation; PD-1
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200mg q3w

SUMMARY:
To investigate whether concurrent Tislelizumab with postoperative chemoradiotherapy would have survival benefit in high Risk HNSCC Patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed squamous cell carcinoma of the head and neck. Site of tumor origin in the oral cavity, oropharynx (p16-), larynx, or hypopharynx
2. With at least one high risk factor after radical surgery ①positive margin; ②close margin（<5mm); ③ENE.
3. No distant metastases
4. No synchronous or concurrent head and neck primary tumors
5. ECOG PS 0-1
6. Adequate organ function including the following:

Absolute neutrophil count (ANC) >= 1.5 * 10^9/l Platelets count >= 80 * 10^9/l Hemoglobin >= 80 g/dl AST and ALT <= 2.5 times institutional upper limit of normal (ULN) Total bilirubin <= 1.5 times institutional ULN Creatinine clearance >30 ml/min 8. Signed written informed consent

Exclusion Criteria:

1. Prior chemotherapy or anti-cancer biologic therapy for any type of cancer, or prior radiotherapy to the head and neck region
2. Other previous cancer, except for in situ cervical cancer and cutaneous basal cell carcinoma
3. Pregnant or breast-feeding females, or females and males of childbearing potential not taking adequate contraceptive measures
4. Uncontrolled concomitant illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
5. Active, known or suspected autoimmune disease such as interstitial pneumonia, uveitis, Crohn's disease, autoimmune thyroiditis. Subjects with cured childhood asthma, type I diabetes mellitus and hypothyroidism only requiring hormone replacement, or skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment
6. Using systemic immunosuppressive agents and continue the dose within 2 weeks prior to the enrollment;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year disease free survival | 1 year
  from date of enrollment until date of first documented disease progression or from date of enrollment until date of first documented disease progression or death from any cause

SECONDARY OUTCOMES:
Overall survival | 2 years
  from date of enrollment until death from any cause
Number of participants with treatment-related acute toxicity as assessed weekly by CTCAE v4.0 during the course of treatment | up to 3 months after completion of radiotherapy
  Acute toxicity profiles, graded according to the NCI CTCAE version 4.0